CLINICAL TRIAL: NCT01970319
Title: Mechanisms and Reversibility of Heart Failure Associated With Diabetes
Acronym: MRHD
Status: Completed | Type: Observational
Sponsor: Dr. Peter Swoboda (Other)
Responsible Party: Sponsor-Investigator, Dr. Peter Swoboda, BHF Clinical Research Training Fellow, University of Leeds
Organization: University of Leeds (Other)
Other Study IDs: 14606
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic with nephropathy
- Diabetics without nephropathy

SUMMARY:
Patients with diabetes have a higher incidence of heart failure and worse outcomes than normoglycaemic subjects. Basic science research has suggested many mechanisms for this observation including endothelial dysfunction, abnormal calcium handling, fibrosis and activation of the renin-angiotensin-aldosterone system (RAAS), but clinical data are lacking. In this study the investigators will investigate the relationship between diabetes and heart failure by exploring the correlation between microvascular dysfunction and cardiac magnetic resonance (CMR) markers of left ventricular (LV) hypertrophy, cardiac dysfunction and fibrosis. The investigators also propose to see if this relationship is independent of blood pressure and markers of RAAS activity. This could have important clinical ramifications in type 2 diabetes by increasing the indications for treatment with RAAS inhibition or making a case for lower blood pressure targets.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

* Known cardiac or renal disease
* Uncontrolled hypertension
* Treatment with ACEi/ARB
* Treatment with insulin
* Contraindication to CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Left ventricle mass | One year

SECONDARY OUTCOMES:
Left ventricle function | 1 year
RAAS activity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

REFERENCES:
- [Derived] Swoboda PP, Erhayiem B, Kan R, McDiarmid AK, Garg P, Musa TA, Dobson LE, Witte KK, Kearney MT, Barth JH, Ajjan R, Greenwood JP, Plein S. Cardiovascular magnetic resonance measures of aortic stiffness in asymptomatic patients with type 2 diabetes: association with glycaemic control and clinical outcomes. Cardiovasc Diabetol. 2018 Mar 5;17(1):35. doi: 10.1186/s12933-018-0681-4. PMID 29506523
- [Derived] Swoboda PP, McDiarmid AK, Erhayiem B, Ripley DP, Dobson LE, Garg P, Musa TA, Witte KK, Kearney MT, Barth JH, Ajjan R, Greenwood JP, Plein S. Diabetes Mellitus, Microalbuminuria, and Subclinical Cardiac Disease: Identification and Monitoring of Individuals at Risk of Heart Failure. J Am Heart Assoc. 2017 Jul 17;6(7):e005539. doi: 10.1161/JAHA.117.005539. PMID 28716801